CLINICAL TRIAL: NCT01407471
Title: Interest of Topical Spironolactone's Administration to Prevent Corticoid-induced Epidermal Atrophy
Acronym: SPIREPI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Société de Dermatologie Française (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P071011
Record Dates: First submitted 2011-06-30; First posted 2011-08-02 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-02

CONDITIONS: Cutaneous Atrophy Due to Corticosteroids
Keywords: aldosterone; clobetasol; atrophy; skin; epidermis; wound healing; mineral corticoid receptor; spironolactone
MeSH Terms: conditions — Atrophy | interventions — Clobetasol; Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Clobetasol + Spironolactone (Experimental): 0.05% clobetasol and 5% spironolactone
  Interventions: Drug: Clobetasol + Spironolactone
- Clobetasol + Placebo (Active Comparator): 0.05% clobetasol + inert excipient
  Interventions: Drug: Clobetasol + Placebo
- Placebo + Spironolactone (Active Comparator): Inert excipient + 5% spironolactone
  Interventions: Drug: Placebo + Spironolactone
- Placebo + placebo (Placebo Comparator): Inert excipient
  Interventions: Drug: Placebo + Placebo

INTERVENTIONS:
Drug: Clobetasol + Spironolactone — One application 6 days a week during 4 weeks
  Arms: Clobetasol + Spironolactone
Drug: Clobetasol + Placebo — One application 6 days a week during 4 weeks
  Arms: Clobetasol + Placebo
Drug: Placebo + Spironolactone — One application 6 days a week during 7 weeks
  Arms: Placebo + Spironolactone
Drug: Placebo + Placebo — One application 6 days a week during 7 weeks
  Arms: Placebo + placebo

SUMMARY:
The purpose of this study is to determine whether spironolactone could significantly reduce cutaneous atrophy due to corticosteroids.

DETAILED DESCRIPTION:
skin cutaneous atrophy due to corticosteroids limits the long-term use of highly potent topical glucocorticoids which are the treatment of choice for many inflammatory skin diseases. This atrophy results in fragile skin, delay of healing, purpura, irreversible striae, telangiectasia and secondary infections. Up to now, no treatments can prevent efficiently skin atrophy.

The mineralocorticoid receptor, belonging to the superfamily of nuclear receptors, is expressed in human epidermis but its actual function is unknown. Experimental results in animals obtained in INSERM unit U772 by Dr N FARMAN suggest that spironolactone which is a mineralocorticoid receptor antagonist 1- might limit epidermal atrophy and 2- might promote healing.

Study description We propose to test clinically these hypotheses for the first time on humans, at the CIC in BICHAT's hospital on healthy volunteers: 1- by applying on the skin a highly potent cutaneous corticosteroids in association or not with spironolactone, 2- by applying or not spironolactone on wounds after 3-mm punch biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers of both sex, aged between 20 and 50 years
* Woman with effective contraception and pregnancy test negative before inclusion.
* Subject considered healthy after a detailed review (interview, clinical examination)
* Subject belonging to a social security scheme (beneficiary or have the right)
* Subject having signed a free and informed consent
* Integrity of the skin at forearms
* Subject available the next 7 weeks and able to go to CIC once a day from Monday to Friday
* Subject accepting four skin biopsies at D29
* no washing forearms during 2 hours after applications

Exclusion Criteria:

* Chronic Alcoholism
* Drug-addiction (comprehensive interview with a sampling in case of doubt)
* Woman pregnant or breast-feeding
* Subject involved in another trial or in exclusion period of another protocol
* Subject has already received more than 3700 Euros in compensation for damages suffered constraints in the past 12 months for his involvement in biomedical researches
* Subject has already participated in this protocol
* Phototypes 5 and 6
* Clinical skin atrophy
* History of severe chronic skin disease
* Problems of healing
* Treatment with oral corticosteroids, mineralocorticoids or spironolactone (Aldactone, Flumach, Practon, Spiroctan, Spironone, Aldactazine, ALDALIX, Practazin, Spiroctazine ...)

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
histological measure of epidermal thickness | day 29
  biopsies will be performed in the center of the treated sites. Epidermal thickness will be measured from the basal lamina to the lower border of the stratum corneum. This will be determined by image analysis from the average of fields per skin section.

SECONDARY OUTCOMES:
delay of healing after skin biopsies performed on day 29 | days 32, 36, 39, 43, 46, 50
Dermis thickness evaluated by ultrasound | days 1, 15, 29
Mineral receptors and glucoreceptors expression ratio performed by immunohistochemistry | day 29

CONTACTS AND LOCATIONS:
Overall Officials: Eve MAUBEC, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Bichat Hospital, Paris, France

REFERENCES:
- [Background] Farman N, Maubec E, Poeggeler B, Klatte JE, Jaisser F, Paus R. The mineralocorticoid receptor as a novel player in skin biology: beyond the renal horizon? Exp Dermatol. 2010 Feb;19(2):100-7. doi: 10.1111/j.1600-0625.2009.01011.x. Epub 2009 Nov 18. PMID 19925636
- [Background] Bayo P, Sanchis A, Bravo A, Cascallana JL, Buder K, Tuckermann J, Schutz G, Perez P. Glucocorticoid receptor is required for skin barrier competence. Endocrinology. 2008 Mar;149(3):1377-88. doi: 10.1210/en.2007-0814. Epub 2007 Nov 26. PMID 18039792
- [Background] Sainte Marie Y, Toulon A, Paus R, Maubec E, Cherfa A, Grossin M, Descamps V, Clemessy M, Gasc JM, Peuchmaur M, Glick A, Farman N, Jaisser F. Targeted skin overexpression of the mineralocorticoid receptor in mice causes epidermal atrophy, premature skin barrier formation, eye abnormalities, and alopecia. Am J Pathol. 2007 Sep;171(3):846-60. doi: 10.2353/ajpath.2007.060991. Epub 2007 Aug 3. PMID 17675581
- [Background] Stojadinovic O, Lee B, Vouthounis C, Vukelic S, Pastar I, Blumenberg M, Brem H, Tomic-Canic M. Novel genomic effects of glucocorticoids in epidermal keratinocytes: inhibition of apoptosis, interferon-gamma pathway, and wound healing along with promotion of terminal differentiation. J Biol Chem. 2007 Feb 9;282(6):4021-34. doi: 10.1074/jbc.M606262200. Epub 2006 Nov 9. PMID 17095510
- [Background] Leyvraz C, Charles RP, Rubera I, Guitard M, Rotman S, Breiden B, Sandhoff K, Hummler E. The epidermal barrier function is dependent on the serine protease CAP1/Prss8. J Cell Biol. 2005 Aug 1;170(3):487-96. doi: 10.1083/jcb.200501038. PMID 16061697
- [Background] List K, Haudenschild CC, Szabo R, Chen W, Wahl SM, Swaim W, Engelholm LH, Behrendt N, Bugge TH. Matriptase/MT-SP1 is required for postnatal survival, epidermal barrier function, hair follicle development, and thymic homeostasis. Oncogene. 2002 May 23;21(23):3765-79. doi: 10.1038/sj.onc.1205502. PMID 12032844
- [Background] Mauro T, Guitard M, Behne M, Oda Y, Crumrine D, Komuves L, Rassner U, Elias PM, Hummler E. The ENaC channel is required for normal epidermal differentiation. J Invest Dermatol. 2002 Apr;118(4):589-94. doi: 10.1046/j.1523-1747.2002.01721.x. PMID 11918703
- [Background] Perez P, Page A, Bravo A, Del Rio M, Gimenez-Conti I, Budunova I, Slaga TJ, Jorcano JL. Altered skin development and impaired proliferative and inflammatory responses in transgenic mice overexpressing the glucocorticoid receptor. FASEB J. 2001 Sep;15(11):2030-2. doi: 10.1096/fj.00-0772fje. Epub 2001 Jul 24. PMID 11511512
- [Background] Brouard M, Casado M, Djelidi S, Barrandon Y, Farman N. Epithelial sodium channel in human epidermal keratinocytes: expression of its subunits and relation to sodium transport and differentiation. J Cell Sci. 1999 Oct;112 ( Pt 19):3343-52. doi: 10.1242/jcs.112.19.3343. PMID 10504339
- [Background] Roudier-Pujol C, Rochat A, Escoubet B, Eugene E, Barrandon Y, Bonvalet JP, Farman N. Differential expression of epithelial sodium channel subunit mRNAs in rat skin. J Cell Sci. 1996 Feb;109 ( Pt 2):379-85. doi: 10.1242/jcs.109.2.379. PMID 8838661
- [Background] Kenouch S, Lombes M, Delahaye F, Eugene E, Bonvalet JP, Farman N. Human skin as target for aldosterone: coexpression of mineralocorticoid receptors and 11 beta-hydroxysteroid dehydrogenase. J Clin Endocrinol Metab. 1994 Nov;79(5):1334-41. doi: 10.1210/jcem.79.5.7962326.
- [Background] Messina M, Manieri C, Musso MC, Pastorino R. Oral and topical spironolactone therapies in skin androgenization. Panminerva Med. 1990 Apr-Jun;32(2):49-55. PMID 2147469
- [Background] Maubec E, Laouenan C, Deschamps L, Nguyen VT, Scheer-Senyarich I, Wackenheim-Jacobs AC, Steff M, Duhamel S, Tubiana S, Brahimi N, Leclerc-Mercier S, Crickx B, Perret C, Aractingi S, Escoubet B, Duval X, Arnaud P, Jaisser F, Mentre F, Farman N. Topical Mineralocorticoid Receptor Blockade Limits Glucocorticoid-Induced Epidermal Atrophy in Human Skin. J Invest Dermatol. 2015 Jul;135(7):1781-1789. doi: 10.1038/jid.2015.44. Epub 2015 Feb 10. PMID 25668238